CLINICAL TRIAL: NCT03534258
Title: Does Use of Rapid Response EEG Impact Clinical Decision Making
Acronym: DECIDE
Status: Completed | Type: Observational
Sponsor: Ceribell Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1825
Record Dates: First submitted 2018-04-19; First posted 2018-05-23 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Nonconvulsive Status Epilepticus; Seizures
MeSH Terms: conditions — Status Epilepticus; Seizures | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Ceribell Rapid Response EEG, Survey — This trial will qualitatively examine how information from rapid response and conventional EEG data changes physicians' diagnostic suspicion or their treatment decisions and confidence levels. In addition, the results will examine the mean time to EEG lead placement, and ease of use.

SUMMARY:
This study is designed as a prospective, non-randomized, observational, multicenter clinical trial. The primary aim of this study is to observe if the use of the rapid responds electroencephalography (EEG) system impacts physician decision making. Secondary aims include exploring the safety and performance information of the Ceribell EEG system compared to conventional EEG system. The study will recruit physicians (Faculty physicians and Trainees) at up to five institutions and examine the impact of rapid response EEG when providing care to patients in whom EEG recording has been ordered for clinical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing clinically ordered EEGs.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve two groups of subjects:
  1. Physicians (faculty and trainees), who will be asked to fill out a nonsensitive questionnaire. These are members of Epilepsy and Neuro-ICU team (attendings, fellows, or residents) who are actively involved in the care of patients and know the patient's history of present illness.
  2. Patients undergoing clinically ordered EEGs.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in physicians' diagnosis decision | through study completion, an average of 1 year
  Physician will record their diagnostic assessment of seizure in Yes or No.
Change in physicians' diagnosis confidence | through study completion, an average of 1 year
  Physician will rate their diagnosis confidence with a score between 1 to 5
Change in physicians' treatment decision | through study completion, an average of 1 year
  Physician will record their treatment decision in Yes or No.
Change in physicians' treatment confidence | through study completion, an average of 1 year
  Physician will rate their treatment confidence with a score between 1 to 5

SECONDARY OUTCOMES:
Time from order to EEG arrival | through study completion, an average of 1 year
  Time from EEG order to EEG arrival will be recorded for both Ceribell EEG and conventional EEG
Set up time | through study completion, an average of 1 year
  Time from EEG arrival to the first EEG recording will be recorded for both Ceribell EEG and conventional EEG
Ease of use | through study completion, an average of 1 year
  Ease of use will be recorded with a score of 1-5
Signal Quality of EEG | through study completion, an average of 1 year
  Signal Quality of Ceribell EEG as measured with Hjorth parameters (Hjorth Activity, Hjorth Mobility, Hjorth Complexity) will be compared to signal quality of conventional EEG acquired from the same patients

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California Los Angeles, Los Angeles, California
  - Rush University Medical Center Pob, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vespa PM, Olson DM, John S, Hobbs KS, Gururangan K, Nie K, Desai MJ, Markert M, Parvizi J, Bleck TP, Hirsch LJ, Westover MB. Evaluating the Clinical Impact of Rapid Response Electroencephalography: The DECIDE Multicenter Prospective Observational Clinical Study. Crit Care Med. 2020 Sep;48(9):1249-1257. doi: 10.1097/CCM.0000000000004428. PMID 32618687